CLINICAL TRIAL: NCT01968551
Title: A Phase 3 Open-Label Study to Evaluate Switching From Optimized Stable Antiretroviral Regimens Containing Darunavir to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Single Tablet Regimen (STR) Plus Darunavir (DRV) in Treatment Experienced HIV-1 Positive Adults
Brief Title: Phase 3 Open-Label Study to Evaluate Switching From Optimized Stable Antiretroviral Regimens Containing Darunavir to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Fixed Dose Combination (FDC) Plus Darunavir (DRV) in Treatment Experienced HIV-1 Positive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-292-0119
Record Dates: First submitted 2013-09-26; First posted 2013-10-24 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2017-07

CONDITIONS: HIV-1; HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: HIV-1; HIV; Treatment-Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants will receive E/C/F/TAF FDC + DRV once daily with food for 48 weeks.
  Based on safety and efficacy data from Cohort 1 at Week 4, the participants will be randomized into Cohort 2. The participants in Cohort 1 will continue receiving E/C/F/TAF FDC + DRV through 48 weeks.
  Interventions: Drug: E/C/F/TAF; Drug: DRV
- Cohort 2, Treatment Group 1 (Experimental): Participants will be randomized to receive E/C/F/TAF FDC+DRV once daily with food for 48 weeks.
  Interventions: Drug: E/C/F/TAF; Drug: DRV
- Cohort 2, Treatment Group 2 (Active Comparator): Participants will be randomized to continue on their baseline DRV-containing ARV regimen for 48 weeks.
  Interventions: Drug: Baseline DRV- containing ARV regimen

INTERVENTIONS:
Drug: E/C/F/TAF — 150/150/200/10 mg FDC tablet administered orally once daily
  Other Names: Genvoya®
  Arms: Cohort 1; Cohort 2, Treatment Group 1
Drug: DRV — 800 mg tablet administered orally once daily
  Arms: Cohort 1; Cohort 2, Treatment Group 1
Drug: Baseline DRV- containing ARV regimen — Participants will take their baseline DRV- containing ARV regimen as prescribed.
  Arms: Cohort 2, Treatment Group 2

SUMMARY:
The primary objective of this study is to evaluate the efficacy of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) fixed dose combination (FDC) plus darunavir (DRV) relative to current antiretroviral regimens (ARV) in virologically suppressed, HIV-1 positive participants with HIV-1 RNA <50 copies/mL at Week 24.

This study consists of 48 weeks of open-label phase followed by an optional Extension Phase in which all the participants will receive E/C/F/TAF+DRV.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and sign a written informed consent form
* History of at least two prior antiretroviral regimens, and history of resistance to at least two different classes of antiretroviral agents
* Plasma HIV-1 RNA levels < 50 copies/mL at screening. Virologically suppressed on the current antiretroviral regimen containing darunavir 600 mg twice a day or 800 mg once daily continuously for ≥ 4 months preceding the screening visit and have maintained documented undetectable plasma HIV-1 RNA levels (< 50 copies/mL) and must have documentation of genotype/phenotype prior to current regimen which shows no darunavir associated resistance mutation.
* Currently receiving raltegravir, elvitegravir, or dolutegravir (50 mg once daily, but not twice daily), or have never received integrase inhibitor, or have documentation of genotype/phenotype within 12 months prior to current regimen which must show no evidence of resistance to integrase inhibitors
* Normal ECG
* Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min according to the Cockcroft Gault formula for creatinine clearance
* Hepatic transaminases (AST and ALT) ≤ 5 × upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function (absolute neutrophil count ≥ 1,000/mm^3; platelets ≥ 50,000/mm^3; hemoglobin ≥ 8.5 g/dL)
* Serum amylase ≤ 5 × ULN (individuals with serum amylase > 5 × ULN will remain eligible if serum lipase is ≤ 5 × ULN)
* A female individual is eligible to enter the study if it is confirmed that she is:

  * Not pregnant or nursing
  * Of non-childbearing potential (i.e., women who have had a hysterectomy, have had both ovaries removed or medically documented ovarian failure, or are postmenopausal women > 54 years of age with cessation (for ≥ 12 months) of previously occurring menses), or
  * Of childbearing potential and agrees to utilize highly effective contraception methods or be non-heterosexually active or practice sexual abstinence from screening throughout the duration of study treatment and for 30 days following the last study drug dose.
  * Female individuals who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing.
* Male individuals must agree to utilize a highly effective method of contraception during heterosexual intercourse or be non-heterosexually active, or practice sexual abstinence from first dose throughout the study period and for 30 days following the last study drug dose.
* Male individuals must agree to refrain from sperm donation from first dose until at least 30 days after the last study drug dose.

Key Exclusion Criteria:

* A new AIDS-defining condition diagnosed within the 30 days prior to screening (except CD4 cell count and/or percentage criteria)
* Hepatitis B surface antigen (HBsAg) positive
* Individuals receiving drug treatment for Hepatitis C, or individuals who are anticipated to receive treatment for Hepatitis C during the course of the study.
* Must not have Q151M, T69ins, or > 3 thymidine analogue mutations (TAMS) present on documented historic genotype report
* Individuals experiencing decompensated cirrhosis
* Females who are breastfeeding
* Positive serum pregnancy test
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance use that may interfere with individual's study compliance
* A history of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma.
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Day 1 visit
* Any other clinical condition or prior therapy that would make the individual unsuitable for the study or unable to comply with dosing requirements
* Participation in any other clinical trial (including observational trials) without prior approval from the sponsor is prohibited while participating in this trial
* Individuals receiving ongoing therapy with any of the disallowed medications, including drugs not to be used with elvitegravir, cobicistat, emtricitabine, TAF, or DRV; or individuals with any known allergies to the study drugs.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2015-07-21 (Actual); Study Completion 2016-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (62):
- United States (56):
  - Pueblo Family Physicians, Ltd., Phoenix, Arizona
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Kaiser Permanente, Hayward, California
  - Long Beach Education and Research Consultants, Long Beach, California
  - Peter J Ruane, MD, Inc., Los Angeles, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - Kaiser San Francisco Division of Research, San Francisco, California
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Gary J.Richmond, MD, P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Valuhealthmd/Idocf, Orlando, Florida
  - Infectious Diseases Associates of NW FL, Pensacola, Florida
  - Hillsborough County Health Department, Tampa, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - AIDS Research and Treatment Center of the Treasure Coast, Vero Beach, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - Atlanta ID Group, Atlanta, Georgia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Mercer University, Mercer Medicine, Macon, Georgia
  - The Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - Johns Hopkins University, Lutherville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Harvard Medical School, Boston, Massachusetts
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - The Kansas City Free Health Clinic/ KC Care Clinic, Kansas City, Missouri
  - Central West Clinical Research, St Louis, Missouri
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Southwest CARE Center, Santa Fe, New Mexico
  - Albany Medical College, Albany, New York
  - New York Hospital Queens, Flushing, New York
  - Beth Israel Medical Center, New York, New York
  - Weill Medical College, New York, New York
  - University of Rochester, Rochester, New York
  - Carolinas Medical Center--Myer's Park, Charlotte, North Carolina
  - Duke University Health System, Durham, North Carolina
  - East Carolina University The Brody School of Medicine, Infectious Diseases, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System CARE Center, Akron, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - North Texas infectious Diseases Consultants, PA, Dallas, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - University of Utah, Salt Lake City, Utah
  - Clinical Alliance for Research & Education - Infectious Diseases (CARE-ID), Annandale, Virginia
  - Peter Shalit, MD, Seattle, Washington
- Canada (6):
  - Southern Alberta Clinic, Calgary, Alberta
  - Vancouver ID Research & Care Centre Society, Vancouver, British Columbia
  - Wrha - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Maple Leaf Research, Toronto, Ontario
  - Clinique médicale L'actuel, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Background] Huhn GD, Tebas P, Gallant J, Wilkin T, Cheng A, Yan M, Zhong L, Callebaut C, Custodio JM, Fordyce MW, Das M, McCallister S. A Randomized, Open-Label Trial to Evaluate Switching to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Plus Darunavir in Treatment-Experienced HIV-1-Infected Adults. J Acquir Immune Defic Syndr. 2017 Feb 1;74(2):193-200. doi: 10.1097/QAI.0000000000001193. PMID 27753684
- [Background] Greg Huhn, Pablo Tebas, Joel Gallant et al. Strategic Simplification: the Efficacy and Safety of Switching to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Plus Darunavir (DRV) in Treatment-Experienced HIV-1-Infected Adults (NCT01968551). IDWeek; 2015 San Diego, CA Oct. 7-11.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and Canada. The first participant was screened on 3 September 2013. The last study visit occurred on 09 July 2016.
Pre-assignment Details: 231 participants were screened.
Groups:
- Cohort 1: E/C/F/TAF+DRV: Open-Label (OL) Phase: Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (Genvoya®; E/C/F/TAF) (150/150/200/10 mg) fixed-dose combination (FDC) tablet plus Darunavir (DRV) (800 mg) tablet administered orally once daily for up to 48 weeks
  Open-Label Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus Darunavir (DRV) (800 mg) tablet administered orally once daily
- Cohort 2: E/C/F/TAF+DRV: Open-Label Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily for up to 48 weeks
  Open-Label Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily
- Cohort 2: Stay on Baseline Regimen (SBR): Open-Label Phase: Participants stayed on their baseline DRV- containing regimen administered according to the prescribing information for up to 48 weeks.
  Open-Label Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily
Period: Open Label Phase (48 Weeks)
Arm/Group | Cohort 1: E/C/F/TAF+DRV | Cohort 2: E/C/F/TAF+DRV | Cohort 2: Stay on Baseline Regimen (SBR)
Started | 22 | 90 | 46
Completed | 20 | 87 | 41
Not Completed | 2 | 3 | 5
Not completed — Randomized but Never Treated | 1 | 1 | 0
Not completed — Investigator's Discretion | 0 | 1 | 0
Not completed — Withdrew Consent | 1 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2
Period: Extension Phase
Arm/Group | Cohort 1: E/C/F/TAF+DRV | Cohort 2: E/C/F/TAF+DRV | Cohort 2: Stay on Baseline Regimen (SBR)
Started | 20 | 87 | 34 (7 participant completed the Open-Label Phase, but did not enter in the Extension Phase)
Completed | 19 | 86 | 30
Not Completed | 1 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Withdrew Consent | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included:
  * Cohort 1: participants who (1) were enrolled into Cohort 1 and (2) received at least 1 dose of study drug during the OL Phase or the Extension Phase
  * Cohort 2: participants who (1) were randomized into Cohort 2 and (2) received at least 1 dose of study drug during the OL Phase or the Extension Phase
Groups:
- Cohort 1: E/C/F/TAF+DRV; Cohort 2: E/C/F/TAF+DRV: Open-Label Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily with food for up to 48 weeks
  Open-Label Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily
- Cohort 2: SBR: Open-Label Phase: Participants stayed on their baseline DRV- containing regimen administered according to the prescribing information for up to 48 weeks
  Open-Label Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily
- Total: Total of all reporting groups
Arm/Group | Cohort 1: E/C/F/TAF+DRV | Cohort 2: E/C/F/TAF+DRV | Cohort 2: SBR | Total
Number analyzed (Participants) | 21 | 89 | 46 | 156
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53 (5.7) | 49 (8.2) | 47 (9.4) | 49 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 16 | 18 | 42
  Male | 13 | 73 | 28 | 114
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Black | 12 | 35 | 26 | 73
  Native Hawaiian or Pacific Islander | 0 | 1 | 0 | 1
  White | 9 | 51 | 17 | 77
  Not Permitted | 0 | 0 | 0 | 0
  Other | 0 | 0 | 3 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 12 | 7 | 21
  Not Hispanic or Latino | 19 | 77 | 39 | 135
  Not Permitted | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 9 | 3 | 12
  United States | 21 | 80 | 43 | 144
HIV-1 RNA Category [Number; unit: participants]
  < 50 copies/mL | 19 | 87 | 46 | 152
  ≥ 50 copies/mL | 2 | 2 | 0 | 4
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 700 (372.5) | 562 (260.8) | 571 (245.2) | 583 (275.9)
CD4 Cell Count Category [Number; unit: participants]
  < 200 cells/µL | 1 | 5 | 1 | 7
  ≥ 200 to < 350 cells/µL | 3 | 15 | 7 | 25
  ≥ 350 cells/µL | 17 | 69 | 38 | 124

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Each Treatment Arm in Cohort 2 With HIV-1 RNA < 50 Copies/mL at Week 24
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Full Analysis Set (FAS) in Cohort 2, included all participants who (1) were randomized to Cohort 2 and (2) received at least 1 dose of study drug during the open-label Phase.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 2: E/C/F/TAF+DRV: Open-Label Phase: E/C/F/TDF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily for up to 48 weeks
  Open-Label Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily
Arm/Group | Cohort 2: E/C/F/TAF+DRV | Cohort 2: Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 89 | 46
percentage of participants | 96.6 | 91.3
Statistical Analysis 1: Comparison: Cohort 2: E/C/F/TAF+DRV vs Cohort 2: Stay on Baseline Regimen (SBR); Test type: Non-Inferiority or Equivalence — Null Hypothesis: In Cohort 2, the group switching to E/C/F/TAF + DRV was at least 12% lower than the group remaining on SBR with respect to percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24. Alternative Hypothesis: In Cohort 2, the group switching to E/C/F/TAF + DRV is less than 12% lower than the group remaining on SBR with respect to the proportion of participants with HIV-1 RNA<50 copies/mL at Week 24; p = 0.23, Fisher Exact; Difference in proportion = 5.3, 95.001% CI 2-sided [-3.4 to 17.4] — Difference in percentages of virologic success and its 95.001% confidence interval (CI) calculation was based on exact method. The exact CI was estimated based on unconditional exact method using 2 inverted 1-sided tests with standardized statistic

2. Secondary Outcome: Percentage of Participants in Each Treatment Arm in Cohort 2 With HIV-1 RNA < 50 Copies/mL at Week 48
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Full Analysis Set included participants who (1) were randomized into Cohort 2 and (2) had received at least one dose of study drug during the OL phase of the study.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 2: Stay on Baseline Regimen (SBR): Open-Label Phase: Participants stayed on their baseline DRV- containing regimen administered according to the prescribing information for up to 48 weeks
  Open-Label Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily
Arm/Group | Cohort 2: E/C/F/TAF+DRV | Cohort 2: Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 89 | 46
percentage of participants | 94.4 | 76.1
Statistical Analysis 1: Comparison: Cohort 2: E/C/F/TAF+DRV vs Cohort 2: Stay on Baseline Regimen (SBR); Test type: Non-Inferiority or Equivalence — Null Hypothesis: In Cohort 2, the group switching to E/C/F/TAF + DRV was at least 12% lower than the group remaining on SBR with respect to percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48. Alternative Hypothesis: In Cohort 2, the group switching to E/C/F/TAF + DRV is less than 12% lower than the group remaining on SBR with respect to the proportion of participants with HIV-1 RNA < 50 copies/mL at Week 48; p = 0.004, Fisher Exact; Difference in proportion = 18.3, 95.001% CI 2-sided [3.5 to 33.0] — Difference in percentages of virologic success and its 95.001% CI were calculated based on exact method. The exact CI was estimated based on unconditional exact method using 2 inverted 1-sided tests with the standardized statistic

3. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline; Week 24
Population: Full Analysis Set (FAS) included participants who (1) were randomized into Cohort 2 and (2) had received at least one dose of study drug during the OL phase of the study. Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Cohort 2: E/C/F/TAF+DRV | Cohort 2: Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 88 | 42
cells/μL | 23 (155.2) | 12 (100.9)

4. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells/μL
Groups:
- Cohort 2: E/C/F/TAF+DRV: Open-Label Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800mg) tablet administered orally once daily for up to 48 weeks
  Open-Label Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily
- Cohort 2: Stay on Baseline Regimen (SBR): Open-Label Phase: Participants stayed on their baseline DRV- containing regimen administered according to the prescribing information for up to 48 weeks.
  Open-Label (OL) Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily
Arm/Group | Cohort 2: E/C/F/TAF+DRV | Cohort 2: Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 85 | 39
cells/μL | 5 (162.6) | 41 (104.2)

ADVERSE EVENTS:
Time Frame: Up to a maximum of 97.4 weeks (duration of exposure: Cohort 1 and Cohort 2 = 48 weeks; All E/C/F/TAF = up to maximum of 97.4 weeks)
Description: Safety Analysis Set included all participants in:
  * Cohort 1: who were enrolled into Cohort 1 and received at least 1 dose of study drug during the open-label Phase
  * Cohort 2: who were randomized into Cohort 2 and received at least 1 dose of study drug during the open-label Phase
  * All E/C/F/TAF: who received at least 1 dose of E/C/F/TAF during the Open-Label Phase or Extension Phase
  For Cohort 1 and Cohort 2, only the adverse events that occurred during the Open-Label Phase are reported.
Groups:
- Cohort 2: SBR: Open-Label Phase: Participants stayed on their baseline DRV- containing regimen administered according to the prescribing information for up to 48 weeks.
  Open-Label Extension Phase: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus DRV (800 mg) tablet administered orally once daily
- All E/C/F/TAF: Open- label or Extension Phase: All participants received E/C/F/TAF.
Arm/Group | Cohort 1: E/C/F/TAF+DRV | Cohort 2: E/C/F/TAF+DRV | Cohort 2: SBR | All E/C/F/TAF
Serious Adverse Events (participants affected / at risk) | 1/21 | 9/89 | 1/46 | 20/144
Other Adverse Events (participants affected / at risk) | 13/21 | 56/89 | 28/46 | 104/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: E/C/F/TAF+DRV (N=21) | Cohort 2: E/C/F/TAF+DRV (N=89) | Cohort 2: SBR (N=46) | All E/C/F/TAF (N=144)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Chest pain (General disorders) | 0 | 1 | 0 | 2
Death (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: E/C/F/TAF+DRV (N=21) | Cohort 2: E/C/F/TAF+DRV (N=89) | Cohort 2: SBR (N=46) | All E/C/F/TAF (N=144)
Abdominal pain (Gastrointestinal disorders) | 0 | 5 | 2 | 6
Constipation (Gastrointestinal disorders) | 0 | 5 | 0 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 4 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 1 | 7
Nausea (Gastrointestinal disorders) | 0 | 5 | 0 | 8
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2 | 10
Fatigue (General disorders) | 0 | 4 | 2 | 8
Acute sinusitis (Infections and infestations) | 4 | 1 | 0 | 9
Bronchitis (Infections and infestations) | 3 | 6 | 1 | 14
Influenza (Infections and infestations) | 0 | 1 | 3 | 3
Nasopharyngitis (Infections and infestations) | 0 | 6 | 2 | 8
Oral candidiasis (Infections and infestations) | 2 | 1 | 0 | 3
Otitis media (Infections and infestations) | 2 | 3 | 0 | 7
Pharyngitis (Infections and infestations) | 0 | 5 | 1 | 7
Sinusitis (Infections and infestations) | 3 | 6 | 4 | 15
Upper respiratory tract infection (Infections and infestations) | 3 | 10 | 2 | 27
Viral upper respiratory tract infection (Infections and infestations) | 1 | 4 | 2 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 11 | 3 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 7
Headache (Nervous system disorders) | 1 | 6 | 0 | 16
Hypoaesthesia (Nervous system disorders) | 2 | 1 | 0 | 4
Depression (Psychiatric disorders) | 2 | 2 | 0 | 8
Insomnia (Psychiatric disorders) | 0 | 4 | 1 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3 | 10
Hypertension (Vascular disorders) | 0 | 4 | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other